CLINICAL TRIAL: NCT06569264
Title: Evaluation of Dentin Graft and I-PRF With and Without Vitamin C for Post-extraction Socket Preservation. A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Dentin Graft and I-PRF With and Without Vitamin C for Post-extraction Socket Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Barwa, principle investigator Noha Barwa Master degree student, faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: noha93
Record Dates: First submitted 2024-08-18; First posted 2024-08-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Socket Preservation
Keywords: Socket preservation; Ridge preservation; Demineralized autogenous dentin graft; i-PRF; vitamin C; ascorbic acid
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar ridge preservation using vitamin C with dentin graft and i-PRF (Experimental): Pure vitamin C will be added and extraction socket will be filled with the corresponding graft material. Adding vitamin C to dentin graft and i-PRF might aid in reducing the dimensional changes and marginal bone loss, since it increases osteoblast proliferation and viability during socket preservation. Layers of osteoblast cell morphology can be seen at day 11 with the presence of 25mM of vitamin C. By adding vitamin C to i-PRF we can add the advantages of improving soft tissue quality as well.
  Interventions: Procedure: Alveolar ridge preservation using vitamin C with dentin graft and i-PRF
- Alveolar ridge preservation using autogenous demineralized denting graft combined with i-PRF. (Active Comparator): Autogenous demineralized dentin graft combined with i-PRF and extraction socket will be filled with the corresponding graft material. This mix provided promising clinical outcomes and considered an ideal bioactive graft material for hard tissue regeneration. Autogenous particulate dentin and platelet rich fibrin mix assist healing and counteract pronounced resorption of alveolar process.It can be used as an excellent autogenous graft material to replace other autogenous graft materials, and has shown an ability to maintain the alveolar ridge dimensions because of its osteo-conductive properties. Moreover, dentin graft is used as a cost-effective grafting material during socket preservation.
  Interventions: Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft and i-PRF

INTERVENTIONS:
Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft and i-PRF — Flapless atraumatic extraction. After thorough mechanical cleaning, the sockets will be rinsed with 5 ml of an aqueous 0.125% chlorhexidine digluconate solution, followed by a 5 ml sterile saline rinse to remove tissue debris from the socket. Followed by inspection of extraction socket integrity, using a William's graduated periodontal probe. Extracted teeth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries or restorations using a high-speed fine finishing stone and saline irrigation. The pulp chamber will be cleaned with sterile endodontic files. Teeth will be ground, using hand bone mill. The (ADDG) particles prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralized then washed twice in saline and dried with sterile gauze. The ADDG will be collected in a sterile plastic syringe. For the preparation of i-PRF, 10 mL of venous blood will be drawn into a PET tube and centrifuged at 700rpm for 3 min.
  Arms: Alveolar ridge preservation using autogenous demineralized denting graft combined with i-PRF.
Procedure: Alveolar ridge preservation using vitamin C with dentin graft and i-PRF — Flapless atraumatic extraction. After thorough mechanical cleaning, the sockets will be rinsed with 5 ml of an aqueous 0.125% chlorhexidine digluconate solution, followed by a 5 ml sterile saline rinse to remove tissue debris from the socket. The ADDG particles will be collected in a sterile plastic syringe. For the preparation of i-PRF, 10 mL of venous blood will be drawn into a sterile PET tube and centrifuged at 700 rpm for 3 minutes. The resulting i-PRF liquid layer will then be aspirated from the top of the tube and transferred into the syringe containing the ADDG particles. 25 mM of pure vitamin C , drawn using a micropipette, will be aspirated into the same syringe containing the ADDG-i-PRF mixture. The combined mixture will then be allowed to set for 10 minutes to produce the sticky ADDG.
  Arms: Alveolar ridge preservation using vitamin C with dentin graft and i-PRF

SUMMARY:
The aim of the study is to evaluate radiographic ridge width change following autogenous demineralized dentin graft (ADDG) and i-PRF addition with and without vitamin C (AA) for post extraction socket preservation.

The main question is:

In patient with non-restorable teeth, does adding vitamin C to dentin graft and i-PRF affect the radiographic ridge width of post extraction sockets?

Intervention group:

Alveolar ridge preservation using vitamin C (AA) with autogenous demineralized dentin graft combined with i-PRF.

Adding vitamin C to dentin graft and i-PRF might aid in reducing the dimensional changes, since it increases osteoblast proliferation and viability during socket preservation. Layers of osteoblast cell morphology can be seen at day 11 with the presence of 25mM of vitamin C. By adding vitamin C to i-PRF we can add the advantages of improving soft tissue quality as well.

Control group:

Alveolar ridge preservation using autogenous demineralized denting graft combined with i-PRF.

Dentin particle can be used as an excellent autogenous graft material to replace other autogenous graft materials, it can be used in socket preservation. as it enhances bone formation, and has shown an ability to maintain the alveolar ridge dimensions because of its osteo-conductive properties. Moreover, dentin graft is used as a cost-effective grafting material during socket preservation.

The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. Flapless and atraumatic tooth extraction will be initiated, Then the sockets will be carefully packed with the allocated graft material that are shaped to match the individual size and contours of each socket. Once the grafts are properly adapted to the sockets, they will be covered with the corresponding graft material, and an absorbable gelatin sponge (gelfoam) will be used for socket and graft material coverage and secured using an internal crisscross knot using 5-0 monofilament polypropylene suture material.

DETAILED DESCRIPTION:
Research objective:

Socket preservation is one of the techniques utilized to maintain bone dimension and minimized post-extraction dimensional changes. Adding vitamin C to dentin graft and i-PRF might aid in reducing the dimensional changes, since it increases osteoblast proliferation and viability during socket preservation. By adding vitamin C with i-PRF we can add the advantages of improving soft tissue quality as well. Layers of osteoblast cell morphology can be seen at day 11 with the presence of 25mM of vitamin C. Moreover, dentin graft is used as a cost-effective grafting material during socket preservation.

l. Inclusion criteria:

* ≥ 18 years of age.
* Single extraction of non-molar teeth with periodontally healthy adjacent teeth.
* Non-contributory medial history.
* Non- restorable teeth indicated for extraction.
* Requiring alveolar preservation after tooth extraction prior to placement of dental implant.
* Participants that are eligible for immediate implantation, yet having factors that are hindering these patients from immediate placement of an implant at the time of extraction (ex: Financial related factors - psychological psychological factors - time related factors).
* Cooperative patients who are willing to commit for 3 months follow up.

II. Exclusion criteria:

* Pregnant female.
* Acute infection at extraction site.
* Systemic conditions affecting healing (e.g., diabetes, medications as bisphosphonates...)
* A participant who had radiotherapy or chemotherapy.
* Psychiatric patient, or with a learning disability, or unable to give consent.

Research Procedure in brief:

The study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry- Cairo University, Egypt. Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology, clinic of the department of Oral surgery and clinic of the department of Endodontics -Cairo University. The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. Rinsing with 0.12% chlorhexidine will be instructed.

Preoperative baseline cone-beam computed tomography (CBCT) scan will be conducted.

In both groups, tooth extraction under local anesthesia with articaine HCL 2%, 1:20,000 epinephrine will be performed. Flapless minimally traumatic extraction will be done using thin periotomes and luxators. After thorough mechanical cleaning, the sockets will be rinsed with 5 ml of an aqueous 0.125% chlorhexidine digluconate solution, followed by a 5 ml sterile saline rinse to remove tissue debris from the socket. This procedure will be repeated three times for each socket. Followed by inspection of extraction socket integrity, using a William's graduated periodontal probe. Then, extracted teeth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries or restorations (if present), using a high-speed fine finishing stone and saline irrigation. The pulp chamber will be cleaned with sterile endodontic files. Subsequently, teeth will be ground, using hand bone mill.

The demineralized autogenous tooth graft (ADDG) particles prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralized then washed twice in saline and dried with sterile gauze.

For i-PRF preparation, blood will be withdrawn in plastic tubes without anticoagulant.

The ADDG particles will be collected in a sterile plastic syringe. For the preparation of i-PRF, 10 mL of venous blood will be drawn into a sterile PET tube and centrifuged at 700 rpm (60 g-force) for 3 minutes. The resulting i-PRF liquid layer will then be aspirated from the top of the tube and transferred into the syringe containing the ADDG particles. For the intervention group 25 mM of pure vitamin C , drawn using a micropipette, will be aspirated into the same syringe containing the ADDG-i-PRF mixture. The combined mixture will then be allowed to set for 10 minutes to produce the sticky ADDG.

The extraction socket will be filled with the corresponding graft material, and an absorbable gelatin sponge (gelfoam) will be used for socket and graft material coverage and secured using an internal crisscross knot using 5-0 monofilament polypropylene suture material.

Postoperative care and follow up:

* Patient will be instructed to abstain from trauma on the operative site, not to interfere with the suture and to avoid hot food or vigorous rinsing.
* The patients will be advised to refrain from brushing at the surgical area for the first day after surgery.
* A soft surgical brush will be dispensed for the cleaning of the surgical area after the initial healing phase during the first 2 weeks post surgically.
* Antibiotics and analgesics will be prescribed for 5 days.
* Patients will be instructed to:

  1. Follow the instructions completely.
  2. Keep up a strict follow-up schedule.
  3. Not to touch the surgical area, with the tongue or fingers.
  4. Do not wear any kind of dental appliances, on or around the surgical site.

The sutures will be removed two weeks after the surgery. A final follow-up visit and CBCT scan will be scheduled for three months postoperatively.

Face to face adherence reminder session will take place to stress the post-operative instructions at the following time intervals:

* 3 days and 7 days post-operatively, for clinical assessment of swelling, wound dehiscence, and other adverse events.
* 2 weeks after the operation for follow up.
* Lastly, 3 months before implant placement.

Radiographs:

Radiographic ridge width change (primary outcome), buccal ridge height (BRH), and lingual ridge height (LRH) (secondary outcomes) will be assessed by an independent examiner (RW) on CBCT scans obtained at baseline and 3 months postoperatively.

Histological analysis:

For both groups (test and control), before the implant insertion, the grafted site is to be exposed and biopsies from all sites will be excised using a trephine cylindrical drill graduated to indicate the depth (from 5 to 18 mm) with abundant irrigation using sterile saline. Immediate preservation of biopsies in a 10% formalin solution, and then sent for histologic analysis to be analyzed.

Justification for Selecting Radiographic Ridge Width as the Primary Outcome and Excluding Implant-Related Confounders.

1. The primary outcome measure has been changed from marginal bone loss (MBL) around dental implants to radiographic ridge width after socket preservation to more accurately isolate and quantify the effect of the socket preservation procedure itself (Avila-Ortiz et al., 2019). The decision is based on the understanding that subsequent implant placement introduces significant confounding variables that can mask the graft's true efficacy. Including implant placement in the evaluation phase can mask or distort the true dimensional effects of socket preservation, because implant surgery itself initiates a separate cascade of bone remodeling events that are independent of the grafting procedure (Hämmerle & Tarnow, 2018)
2. Placement of an implant introduces several biological and mechanical factors that can mask or override the dimensional benefits achieved through socket preservation, making it difficult to accurately evaluate the true effect of the graft (Capelli, 2013; Huang et al., 2023) (Hämmerle & Tarnow, 2018).
3. The implant osteotomy itself causes mechanical and thermal trauma, initiating a new remodeling cycle that includes necrosis and resorption of the traumatized bone around the implant surface (Peker Tekdal et al., 2016; Li et al., 2020; Ruiz García et al., 2021), consistent with the classic saucerization described by Wilderman et al. and the broader bone remodeling mechanisms associated with implant placement (Capelli, 2013).
4. Additionally, primary stability and insertion torque produce compression and strain in peri-implant bone, influencing remodeling patterns (Schnitman et al., 2014; Huang et al., 2023).
5. Subsequent functional loading further drives adaptive bone modeling/remodeling based on load distribution (Wiskott et al., 2008; da Silva Mello et al., 2018), including vertical bone formation influenced by mechanical stimulus (Hsieh & Turner, 2001; Robling & Turner, 2009; Anitua et al., 2024).
6. Early peri-implant bone changes are also shaped by biologic width establishment, microgap-associated inflammation, and soft-tissue thickness considerations (Rezaei Esfahrood et al., 2016; Berglundh, 1996; Linkevicius et al., 2018; Puisys et al., 2024; Hämmerle et al.). Prosthetic factors such as abutment height, emergence profile, and prosthetic design further influence marginal bone stability, adding variability unrelated to the original graft (Izzetti et al., 2025; Linkevicius et al., 2010; Linkevicius et al., 2015).
7. Likewise, differences in implant macrodesign, surgical technique, loading protocols, cement management, and soft-tissue biotype contribute additional heterogeneity in crestal bone outcomes (Trombelli et al., 2024; Kreve, 2024; Iorio-Siciliano et al., 2024; Costa et al., 2012; Serino & Ström, 2009; Lang & Berglundh, 2011; Valantijiene et al., 2023; Wilson Jr, 2009; Renvert et al., 2014; Tal et al., 2001; Stoilov et al., 2023).
8. Because all of these factors alter bone after implant placement, the radiographic bone levels measured post-implant represent a mixture of socket-preservation outcomes plus implant-induced remodeling, not the preservation effect alone (Amer et al., 2025; Tomlin et al., 2014).
9. This explains why systematic reviews have shown that although ARP significantly reduces ridge shrinkage, its impact on implant survival and marginal bone levels remains inconclusive (Avila-Ortiz et al., 2019; Vignoletti et al., 2012; Crespi et al., 10-year follow-up study). In summary, once an implant is placed, the implant-not the graft-becomes the dominant determinant of bone remodeling (Capelli, 2013), which can conceal or dilute the measurable benefit of socket preservation.

This study uses a 3-month post-extraction evaluation point to accurately capture the direct biological effect of socket preservation prior to any implant-related remodeling.

The decision to shorten follow-up duration from 6 months to 3 months is supported by:

1. Ridge dimensional changes after tooth extraction occur predominantly within the first 8-12 weeks, as clinical and histologic studies demonstrate that the majority of horizontal and vertical alveolar bone remodeling happens during this early healing phase (Avila-Ortiz et al., 2019; Avila-Ortiz, Couso-Queiruga & Chambrone, 2025). Avila-Ortiz et al. (2019) reported that approximately two-thirds of post-extraction horizontal bone loss, averaging 3.87 mm, occur within the first three months, highlighting the importance of early assessment.
2. Systematic reviews also indicate that the primary benefits of alveolar ridge preservation (ARP) and alveolar ridge reconstruction (ARR) are observed in the very short term, which explains the scarcity of long-term evidence beyond five years (Avila-Ortiz, 2014; Avila-Ortiz, Chambrone & Vignoletti, 2025).
3. Measuring ridge dimensions at 3 months provides a direct evaluation of the biological effect of socket preservation, without confounding by implant-related remodeling caused by surgical trauma, prosthetic loading, or biologic width establishment (Barone et al., 2017; Schropp et al., 2003).
4. Schropp et al. demonstrated that while total ridge width loss at one year averaged 6.1 mm, two-thirds of this loss occurred within the first three months, and changes from 3 to 12 months were minimal. Later timepoints introduce confounding factors, including functional loading and prosthetic procedures, which can obscure the graft effect, and
5. Kotsakis et al. (2023) found no significant difference in ridge width or height between 4-month and 12-month assessments after ARP once baseline was controlled, with no significant difference in alveolar ridge width and height change between the two timepoints, suggesting that dimensional changes occur early and stabilize; these results provide both patients and clinicians more freedom in decision-making regarding implant placement timing.
6. Experimental studies comparing grafted extraction sites evaluated at 8-10 weeks versus 18-20 weeks confirm that ridge dimensions are largely stabilized by the earlier timepoint, even though bone maturation continues (Whetman & Mealey, 2016).
7. A 3-month endpoint also reduces participant burden and cumulative radiation exposure, particularly when using CBCT imaging, in alignment with the ethical principle from the Declaration of Helsinki that research procedures must minimize risk and burden to participants (Association, 2025).
8. Therefore, assessing alveolar ridge width at 3 months after socket preservation ensures construct validity, isolates the true biological effect of the graft, and avoids the confounding influences of implant placement or later remodeling (Avila-Ortiz et al., 2019; Vignoletti et al., 2012

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* ≥ 18 years of age.
* Single extraction of non-molar teeth with periodontally healthy adjacent teeth.
* Non-contributory medial history.
* Non- restorable teeth indicated for extraction.
* Requiring alveolar preservation after tooth extraction prior to placement of dental implant.
* Participants that are eligible for immediate implantation, yet having factors that are hindering these patients from immediate placement of an implant at the time of extraction (ex: Financial related factors - psychological psychological factors - time related factors).
* Cooperative patients who are willing to commit for 3 months follow up.

Exclusion Criteria:

* Pregnant female.
* Acute infection at extraction site.
* Systemic conditions affecting healing (e.g., diabetes, medications as bisphosphonates...)
* A participant who had radiotherapy or chemotherapy.
* Psychiatric patient, or with a learning disability, or unable to give consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Radiographic ridge width change | 3 months
  To ensure the primary outcome directly reflects the biological effect of socket preservation and to avoid confounding introduced by implant surgery and loading, the primary outcome has been refined to radiographic horizontal ridge width change measured at baseline and follow-up timepoints.
  The difference from baseline to 3 months follow-up in the radiographic bucco palatal ridge width.
  CBCT scans will be performed at baseline and 3 months postoperatively. Measurements will be taken at both time points using identical reference points and lines measured at a level of 2 mm below the most coronal cross section and perpendicular to the vertical reference line

SECONDARY OUTCOMES:
Buccal ridge height | 3 months
  CBCT scans will be performed at baseline and 3 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point.The height of the alveolus will be measured at the midbuccal aspect (BH)
Lingual ridge height | 3 months
  CBCT scans will be performed at baseline and 3 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point.The height of the alveolus will be measured at the midlingual aspect (LH).
Percentage of newly formed bone | after 3 months postoperatively.
  Histomorphometric analysis will be performed by quantifying the area percentage occupied by bone, graft particles, and soft tissue stroma relative to the total examined histological area using image analyzer software. The image analyzer will be calibrated to automatically convert the measurement units (pixels) produced by the image analyzer program into actual micrometer units. In both groups, the area percentage of newly formed bone will be estimated in three successive regions of the defect, where region two represented the center of the biopsy, using a magnification of x100.
Histological evaluation of residual graft in human biopsies | after 3 months postoperatively.
  eight bone biopsies will be obtained 3 months following engraftment. During implant placement in grafted sites, trephine bur with an outer diameter of 3.3mm, an inner diameter of 2.8mm and a depth of 6-8mm will be used. The biopsies will be stored in 10% formalin solution, decalcified in EDTA for four weeks, processed and embedded in paraffin forming tissue blocks. The paraffin blocks will be cut longitudinally into sections of 5μm thickness will be cut from the paraffin blocks and stained using hematoxylinand eosin (H&E) or Masson's trichromatic (MT) stains for histological evaluation and histomorphometric analysis. Photomicrographs will be taken using a digital light microscope.
postoperative pain | 2 weeks, 1 month and 3 months
  Visual analogue scale (0-10) 10 is the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Karim fawzy, Professor, Study Director — Cairo University; Nesma Shemais, Lecturer, Study Chair — Cairo University; Noha Barwa, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt